CLINICAL TRIAL: NCT03096314
Title: Vitamin D to Improve Outcomes by Leveraging Early Treatment
Acronym: VIOLET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Boyd Taylor Thompson, Co-Prinicipal Investigator PETAL CCC, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PETAL02VIOLET; 1U01HL123009 (NIH)
Record Dates: First submitted 2017-02-21; First posted 2017-03-30 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Acute Respiratory Distress Syndrome; Vitamin D Deficiency; Critical Illness
Keywords: ARDS; Vitamin D
MeSH Terms: conditions — Respiratory Distress Syndrome; Vitamin D Deficiency; Critical Illness | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High dose vitamin D formulation (Active Comparator): A single dose of 540,000 IU vitamin D3 will be administered within 2 hours of randomization time.
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): A single, liquid enteral placebo dose administered either orally or via naso/orogastric tube will be administered within 2 hours of randomization time.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — 540,000 IU vitamin D3 delivered as a single, liquid enteral dose administered either orally or via naso/orogastric tube
  Other Names: cholecalciferol
  Arms: High dose vitamin D formulation
Drug: Placebo — A single, liquid enteral dose identical in appearance and consistency to cholecalciferol administered either orally or via naso/orogastric tube.
  Arms: Placebo

SUMMARY:
Vitamin D deficiency is a common, potentially reversible contributor to morbidity and mortality among critically ill patients. We conducted a randomized, double-blind, placebo-controlled, phase 3 trial of early vitamin D3 supplementation in critically ill, vitamin D-deficient patients who were at high risk for death. Patients screened as vitamin D deficient (<20 ng/mL) were randomized. Randomization occurred within 12 hours after the decision to admit the patient to an intensive care unit. Eligible patients received a single enteral dose of 540,000 IU of vitamin D3 or matched placebo. The primary end point was 90-day all-cause, all-location mortality.

DETAILED DESCRIPTION:
Primary Objective: To assess the efficacy and safety of early administration of vitamin D3 (cholecalciferol) in reducing mortality and morbidity for vitamin D deficient patients at high risk for Acute Respiratory Distress Syndrome (ARDS) and mortality.

Primary Hypothesis: Early administration of vitamin D3 (cholecalciferol) will improve all-cause, all-location mortality to day 90 in vitamin D deficient patients at high risk for ARDS and mortality.

Methods: Patients were recruited from the emergency departments (EDs), hospital wards, operating rooms, intensive care unites (ICUs) and other acute care areas of the participating PETAL Network Clinical Centers. Screening included a test for Vitamin D (25OHD) levels using either the hospital's clinical laboratory or an FDA-approved point-of-care device (FastPack IP, Qualigen Inc). Patients screened as vitamin D deficient (<20 ng/mL) were randomized. Half of the randomized patients received an early administration of high-dose vitamin D3 and the other half received a placebo. Both active and placebo products were given orally or via naso/orogastric tube.

Rational: Vitamin D has pleiotropic roles in regulating immune function and maintaining epithelial surface integrity. Strong preclinical data support the protective role of vitamin D in regulating pulmonary inflammation and disruption of the alveolar-capillary membrane that are fundamental to ARDS pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Intention to admit to ICU from emergency department, hospital ward, operating room, or outside facility
3. One or more of the following acute risk factors for ARDS and mortality contributing directly to the need for ICU admission:

   Pulmonary
   1. Pneumonia
   2. Aspiration
   3. Smoke Inhalation
   4. Lung contusion
   5. Mechanical ventilation for acute hypoxemic or hypercarbic respiratory failure Extra-Pulmonary
   6. Shock
   7. Sepsis
   8. Pancreatitis
4. Vitamin D deficiency (screening 25OHD level <20 ng/mL)

Exclusion Criteria:

1. Inability to obtain informed consent
2. Unable to randomize within 12 hours of ICU admission decision
3. Unable to take study medication by mouth or enteral tube
4. Baseline serum calcium >10.2 mg/dL (2.54 mmol/L) or ionized calcium >5.2 mg/dL (1.30 mmol/L)
5. Known kidney stone in past year or history of multiple (>1) prior kidney stone episodes
6. Decision to withhold or withdraw life-sustaining treatment (patients are still eligible if they are committed to full support except cardiopulmonary resuscitation if a cardiac arrest occurs)
7. Expect <48 hour survival
8. If no other risk factors present, a) mechanical ventilation primarily for airway protection, pain/agitation control, or procedure; or b) elective surgical patients with routine postoperative mechanical ventilation; or c) anticipated mechanical ventilation duration <24 hours; or d) chronic/home mechanical ventilation for chronic lung or neuromuscular disease (non-invasive ventilation used solely for sleep-disordered breathing is not an exclusion).
9. Prisoner
10. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1358 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boyd Taylor Thompson, MD, Principal Investigator — Massachusetts General Hospital
Locations (47):
- United States (47):
  - UCSF Fresno, Fresno, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - St. Joseph Hospital, Del Norte, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - St. Vincent's Hospital, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mt. Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Akron City Hospital, Akron, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OSU Hospital East Campus, Columbus, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Presbyterian/Mercy/Shadyside, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Swedish Hospital Cherry Hill, Seattle, Washington
  - Swedish Hospital First Hill, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected electronically and stored at the Clinical Coordinating Center at Massachusetts General Hospital (MGH). A de-identified database of all data will be available for use 3 years after the primary publication. Data can be accessed at that point via the National Heart Lung Blood Institute (NHLBI) BioLINCC data and biospecimen repository.

REFERENCES:
- [Derived] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Ginde AA, Brower RG, Caterino JM, Finck L, Banner-Goodspeed VM, Grissom CK, Hayden D, Hough CL, Hyzy RC, Khan A, Levitt JE, Park PK, Ringwood N, Rivers EP, Self WH, Shapiro NI, Thompson BT, Yealy DM, Talmor D. Early High-Dose Vitamin D3 for Critically Ill, Vitamin D-Deficient Patients. N Engl J Med. 2019 Dec 26;381(26):2529-2540. doi: 10.1056/NEJMoa1911124. Epub 2019 Dec 11. PMID 31826336
- See also: Website for the PETAL Network — http://petalnet.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After initial study screening, eligible patients were consented and received secondary screening for vitamin D deficiency; performed via an FDA-approved test (either hospital clinical laboratory or the FastPack IP device (Qualigen Inc., Carlsbad, CA). Participants with a screening 25OHD level <20 ng/mL were randomized for treatment assignment.
Groups:
- High Dose Vitamin D Formulation: Patients at high risk for ARDS and mortality with initial screening 25OHD levels < 20 ng/mL randomized to receive 540,00 IU vitamin D3 (cholecalciferol) as a single, liquid enteral dose, administered either orally or via naso/orogastric tube within 2 hours of randomization.
- Placebo: Patients at high risk for ARDS and mortality with initial screening 25OHD levels < 20 ng/mL randomized to receive placebo (similar in appearance to the vitamin D3 treatment) as a single, liquid enteral dose, administered either orally or via naso/orogastric tube within 2 hours of randomization.
Period: Screened Vitamin D Deficient
Arm/Group | High Dose Vitamin D Formulation | Placebo
Started | 690 | 668 (2 randomized but not included in analysis; 1 treated but inadequate consent and 1 withdrew.)
Completed | 681 | 656
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 9 | 12
Period: Confirmed Vitamin D Deficient
Arm/Group | High Dose Vitamin D Formulation | Placebo
Started | 538 (Confirmed deficient (a prior primary analysis subgroup) is a subgroup of the screened deficient.) | 540 (Confirmed deficient (a prior primary analysis subgroup) is a subgroup of the screened deficient.)
Completed | 531 | 528
Not Completed | 7 | 12

BASELINE CHARACTERISTICS:
Population: There were 1360 patients who screened as vitamin D deficient (all randomized) and received a confirmatory LC/MS/MS test (liquid chromatography tandem mass spectrometry). Subjects with a 25OHD result <20 ng/L by LC/MS/MS were the confirmed deficient cohort and included in the primary analysis (N= 538 in Vit D Arm and N = 540 in Placebo arm).
Groups:
- High Dose Vitamin D Formulation: A single dose of 540,000 IU vitamin D3 will be administered within 2 hours of randomization time.
  Vitamin D3: 540,000 IU vitamin D3
- Placebo: A single, liquid enteral placebo dose administered either orally or via naso/orogastric tube will be administered within 2 hours of randomization time.
  Placebo: A single, liquid enteral dose administered either orally or via naso/orogastric tube
- Total: Total of all reporting groups
Arm/Group | High Dose Vitamin D Formulation | Placebo | Total
Number analyzed (Participants) | 538 | 540 | 1078
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 368 | 379 | 747
  >=65 years | 169 | 161 | 330
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 238 | 467
  Male | 309 | 302 | 611
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 280 | 287 | 567
  Race/Ethnicity: Black | 130 | 122 | 252
  Race/Ethnicity: Non-Black Hispanic | 33 | 31 | 64
  Race/Ethnicity: Other | 15 | 12 | 27
  Race/Ethnicity: Not Available | 80 | 88 | 168
Region of Enrollment [Number; unit: participants]
  United States | 538 | 540 | 1078
Facility residence prior to hospitalization (%) [Count of Participants; unit: Participants] | 33 | 35 | 68
Health-related quality of life by EuroQol (EQ-5D-5L) [Mean (Standard Deviation); unit: score] — The questionnaire provides a simple descriptive profile of a respondent's health state. Index ranges from -0.11 to 1.00 (higher scores are better; 1.00 is perfect health)
  score | 0.7 (0.3) | 0.7 (0.3) | 0.7 (0.3)
Charlson co-morbidity index [Mean (Standard Deviation); unit: index] — The Charlson comorbidity index predicts the one-year mortality for a patient who may have a range of comorbid conditions, such as heart disease, AIDS, or cancer (a total of 22 conditions). Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. Index scores range from 0 to 37, with higher scores indicating more coexisting conditions.
  index | 4.0 (2.9) | 3.5 (6.5) | 3.7 (2.9)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Data missing on some subjects prevented calculating index on total cohort.
  kg/m^2
    number analyzed (Participants) | 524 | 529 | 1053
    (all) | 29.8 (10.1) | 31.0 (11.4) | 30.4 (10.8)
Lung Injury risk factors number (%) [Count of Participants; unit: Participants] — Subjects may have more than one risk factor
  Participants
    Pneumonia | 204 | 181 | 385
    Shock | 192 | 197 | 389
    Sepsis | 185 | 174 | 359
    mechanical ventilation for acute resp failure | 119 | 121 | 240
    Aspiration | 27 | 35 | 62
    Lung contusion | 15 | 18 | 33
    Pancreatitis | 17 | 19 | 36
Medical intensive care unit admission - (%) [Count of Participants; unit: Participants] | 447 | 462 | 909
Total Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: score] — The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems. The score is calculated on admission and every 24 hours until discharge using the worst parameters measured during the prior 24 hours. The score ranges from 0-24; a higher score indicates greater predicted mortality.
  score | 4.1 (2.9) | 4.0 (3.1) | 4 (3)
Lung injury prediction score (LIPS) [Mean (Standard Deviation); unit: score] — The lung injury prediction score (LIPS) is a validated prediction model that uses clinical data at the time of presentation to the emergency department (ED) to identify patients at high risk for ARDS. The score is a sum of 19 components, each of which is assigned points. A score of zero = no lung injury. Missing values are given a value of zero. The score ranges from 0 to 36, with higher scores indicating a higher risk of lung injury (as described in Gajic AJRCCM 2020; PMID 20802164).
  score | 5.3 (2.9) | 5.3 (3.1) | 5.3 (3)
Mechanical Ventilation (%) [Count of Participants; unit: Participants] | 173 | 184 | 357
ARDS (%) [Count of Participants; unit: Participants] | 44 | 44 | 88
Vasopressor use at baseline (%) [Count of Participants; unit: Participants] | 169 | 177 | 346
Vitamin D supplement use in past week (%) [Count of Participants; unit: Participants] | 31 | 24 | 55
Multivitamin use in past week (%) [Count of Participants; unit: Participants] | 38 | 37 | 75
Estimated average daily vitamin D dose [Mean (Standard Deviation); unit: IU] — Population: This variable was analyzed in those participants that received a multivitamin/supplement within 30 days prior to current study hospitalization.
  IU
    number analyzed (Participants) | 57 | 54 | 111
    (all) | 3269 (13118) | 4252 (15094) | 3747.1 (14057.7)
25-hydroxyvitamin D [Mean (Standard Deviation); unit: ng/mL] | 11.2 (4.8) | 11 (4.7) | 11.1 (4.7)
Total serum calcium (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Population: This outcome was analyzed in participants in the confirmed deficient cohort with available serum calcium levels.
  mg/dL
    number analyzed (Participants) | 528 | 526 | 1054
    (all) | 8.3 (0.9) | 8.3 (0.9) | 8.3 (0.9)
Ionized calcium (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Population: This outcome was analyzed in participants in the confirmed deficient cohort with available ionized calcium levels.
  mg/dL
    number analyzed (Participants) | 210 | 212 | 422
    (all) | 4.3 (1.4) | 4.3 (0.9) | 4.3 (1.2)
Creatinine (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Population: This outcome was analyzed in participants in the confirmed deficient cohort with available serum creatinine levels.
  mg/dL
    number analyzed (Participants) | 535 | 539 | 1074
    (all) | 2.2 (2.3) | 2.0 (2.0) | 2.1 (2.2)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: ml/min/1.73m2] — The estimated glomerular filtration rate was calculated based on the following variables: race, sex, and serum creatinine using the formula: CFR = 166 x (Scr/0.7) -0.329 x (0.993) Age. Population: This variable was analyzed in participants in the confirmed deficient cohort and calculated based on available data.
  ml/min/1.73m2
    number analyzed (Participants) | 535 | 539 | 1074
    (all) | 60 (39.3) | 60.9 (36.9) | 60.5 (38.1)

OUTCOME MEASURES:

1. Primary Outcome: All-cause, All-location Mortality to Day 90
Description: Vital status of the patient at day 90 was determined using any of the following methods: medical record review, phone calls to patient, proxy or healthcare facility, review of obituaries, or information from the Centers for Disease Control and Prevention's National Death Index (NDI).
Time Frame: 90 days after randomization
Population: The primary analysis included subjects who had confirmed vitamin D deficiency by LC/MS/MS testing.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 531 | 528
Participants | 125 | 109
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; p = 0.26, Generalized linear model

2. Secondary Outcome: All-cause, All Location Mortality to Day 28
Description: This variable was calculated in participants who were reported alive at day 28. Vital status of the patient at day 28 was determined using any of the following methods: medical record review, phone calls to patient, proxy or healthcare facility, or review of obituaries.
Time Frame: Up to 28 days after randomization
Measure: Number; unit: participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 531 | 528
participants | 92 | 69
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Risk Difference (RD) = 4.3, 95% CI 2-sided [-0.1 to 8.6]

3. Secondary Outcome: Hospital Mortality to Day 90
Description: Analysis of the number of participants who died prior to hospital discharge up to study day 90.
Time Frame: Up to 90 days after randomization
Population: Participant count is based on available data.
Measure: Number; unit: participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 538 | 539
participants | 92 | 72
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Risk Difference (RD) = 3.7, 95% CI 2-sided [-0.5 to 8.0]

4. Secondary Outcome: Alive and Home (Prior Level of Care) at Day 90
Description: This endpoint is the count of participants who have survived and are present at home, defined as pre-hospitalization level of care, at day 90.
Time Frame: 90 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 528 | 526
Participants | 348 | 345
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Risk Difference (RD) = 0.3, 95% CI 2-sided [-5.4 to 6.0]

5. Secondary Outcome: Hospital Length of Stay to Day 90
Description: Number of days from enrollment to the day of study hospital discharge up to day 90. Only calculated for patients that survived through day 90.
Time Frame: 90 days after randomization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 406 | 418
days | 9.1 (9.2) | 10.4 (11.0)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.7 to 0.0]

6. Secondary Outcome: Healthcare Facility Length of Stay to Day 90
Description: Healthcare facility length of stay is the time spent in another hospital or healthcare facility (e.g. long-term acute care [LTAC] hospitals or acute rehabilitation/skilled nursing facility), for the subgroup of participants that were discharged to another healthcare facility after the initial hospitalization. This measure is defined as the number of days from initial hospital discharge to the first facility discharge to home (pre-hospitalization level of care) up to day 90. Healthcare facility LOS is zero for patients discharged to home (pre-hospitalization level of care) from the study hospital. This endpoint will be analyzed only in survivors using SACE methods because healthcare facility length of stay in those who die during the follow-up period is non-informative for this endpoint.
Time Frame: 90 days after randomization
Population: This outcome was analyzed only in survivors using SACE methods because healthcare facility length of stay in those who die during the follow-up period is non-informative for this endpoint.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 402 | 416
days | 6.0 (17.5) | 8.1 (20.4)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-4.8 to 0.4]

7. Secondary Outcome: Ventilator-free Days (VFDs) to Day 28
Description: In participants who survive 28 days, ventilator free days (VFDs) is defined as 28 minus duration of ventilation. Duration of ventilation is counted from the first study day of assisted breathing through the last day of assisted breathing provided the last day is prior to day 28. Or it is counted from the first study day of assisted breathing through day 28. For participants discharged with assisted ventilation prior to day 28, a phone call will be required to assess ventilator status at day 28. Participants discharged prior to day 28 (but not to home) on unassisted breathing will be assumed to remain on unassisted breathing through day 28. Isolated periods of ventilation briefer than 24 hours for surgical procedures and ventilation solely for sleep disordered breathing do not count towards duration of ventilation. In participants who never require assisted breathing, duration of ventilation is zero. Participants who do not survive 28 days will be assigned zero VFD.
Time Frame: 28 days after randomization
Population: Excludes subjects who never required assisted breathing or who did not survive 28 days (considered zero vent free days).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 523 | 534
days | 21.3 (11.3) | 22.1 (10.5)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.1 to 0.5]

8. Secondary Outcome: Health-related Quality of Life by EuroQol (EQ-5D-5L)
Description: Changes in Quality of life score by EuroQol from baseline to day 90. Change was calculated as the value at day 90 minus the value at baseline. The EuroQol score is based on 5 dimensions of perceived problems: Mobility, Self-Care, Anxiety/Depression, Pain/discomfort, and Usual Activities. Problems with each area are assigned a level from 1-5 with level 1 being no problem and level 5 indicating extreme problems. A unique health state score is defined by combining 1 level from each of the 5 dimensions. Responses can be used to calculate a health utility score55 associated with the given health state that ranges from -0.11 to 1.00 (higher scores are better; 1.00 is perfect health).
Time Frame: baseline to study day 90
Population: Subjects alive and able to be contacted at study day 90 and who had a baseline EQ-5D-5L assessment were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 340 | 346
score on a scale | 0.0 (0.2) | -0.0 (0.2)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 0, 95% CI 2-sided [0 to 0.1]

9. Secondary Outcome: Number of Participants Who Developed (New) ARDS to Day 7
Description: Presence of ARDS determined using the PaO2/FiO2 ratio or SpO2/FiO2 ratio (i.e., imputed P/F ratio) and chest x-ray confirmation. PaO2 = partial pressure of arterial oxygen; FiO2 = percentage of inspired oxygen; SpO2 = peripheral capillary oxygen saturation, an estimate of the amount of oxygen in the blood. For participants with P/F <300 or imputed P/F <300, FiO2 ≥40%, and PEEP ≥5 cm H2O, we determined if hypoxemia was valid, acute, and not fully explained by congestive heart failure (CHF) or fluid overload. PEEP = positive end expiatory pressure.
Time Frame: Up to 7 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 411 | 412
Participants | 20 | 17
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Risk Difference (RD) = 0.7, 95% CI 2-sided [-2.1 to 3.6]

10. Secondary Outcome: Severity of Acute Respiratory Distress Syndrome (ARDS)
Description: Severity of ARDS is determined using the PaO2/FiO2 ratio or SpO2/FiO2 ratio and confirmation of ARDS through chest x-ray reviews. The breakout of mild to severe was categorized as P/F or imputed P/F ratio of 201-300 (mild), 100-200 (moderate), or less than 100 (severe). This physiologic outcome is one of three key organ systems (respiratory, renal, and cardiovascular) used to assess change in organ failure severity from randomization up to study day 7.
Time Frame: 7 days after randomization
Population: Those subjects that developed new ARDS after randomization were analyzed for severity.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 20 | 17
Participants
  Mild | 6 | 4
  Moderate | 9 | 12
  Severe | 5 | 1
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Mild ARDS; Test type: Superiority; Risk Difference (RD) = 6.5, 95% CI 2-sided [-22.0 to 34.9]
Statistical Analysis 2: Comparison: High Dose Vitamin D Formulation vs Placebo; Moderate ARDS; Test type: Superiority; Risk Difference (RD) = -25.6, 95% CI 2-sided [-56.3 to 5.1]
Statistical Analysis 3: Comparison: High Dose Vitamin D Formulation vs Placebo; Severe ARDS; Test type: Superiority; Risk Difference (RD) = 19.1, 95% CI 2-sided [-2.9 to 41.1]

11. Secondary Outcome: Worst Acute Kidney Injury (AKI)
Description: This physiologic outcome is one of three key organ systems (respiratory, renal, and cardiovascular) used to assess change in organ failure severity from randomization up to study day 7. Worst AKI was determined by using highest daily creatinine values or new use of dialysis/ renal replacement therapy (chronic dialysis participants were excluded). Mild: On-study creatinine levels 1.5 times greater than baseline value or 0.3 mg/dL over the prehospital value. Moderate: On-study creatinine levels 2 times greater than the baseline pre-hospital value. Severe: On-study creatinine creatinine levels are 3 times greater than baseline prehospital value, or the on-study creatinine level is over 4 mg/dL with an acute (1 day) 0.5 mg/dL rise, or participant is on new renal replacement therapy.
Time Frame: Up to 7 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 484 | 495
Participants
  None | 285 | 297
  Mild | 70 | 77
  Moderate | 48 | 52
  Severe | 81 | 69
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; No AKI; Test type: Superiority; Risk Difference (RD) = -1.1, 95% CI 2-sided [-7.3 to 5.0]
Statistical Analysis 2: Comparison: High Dose Vitamin D Formulation vs Placebo; Mild AKI; Test type: Superiority; Risk Difference (RD) = -1.1, 95% CI 2-sided [-5.6 to 3.4]
Statistical Analysis 3: Comparison: High Dose Vitamin D Formulation vs Placebo; Moderate AKI; Test type: Superiority; Risk Difference (RD) = -0.6, 95% CI 2-sided [-4.4 to 3.2]
Statistical Analysis 4: Comparison: High Dose Vitamin D Formulation vs Placebo; Severe AKI; Test type: Superiority; Risk Difference (RD) = 2.8, 95% CI 2-sided [-1.7 to 7.3]

12. Secondary Outcome: New Renal Replacement Therapy (RRT)
Description: Participants who were on chronic dialysis at baseline were excluded from the analysis. Participants who started renal replacement therapy on a study day after day 0 and inclusive of day 7 were considered as having new renal replacement therapy. Those who have never started renal replacement therapy over days 0-7 were considered as not having new renal replacement therapy.
Time Frame: Up to 7 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 489 | 500
Participants | 20 | 18
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Risk Difference (RD) = 0.5, 95% CI 2-sided [-1.9 to 2.9]

13. Secondary Outcome: Highest Creatinine Levels
Description: The highest recorded creatinine values is taken from available levels reported across the 7 study days for each patient.
Time Frame: Up to 7 days after randomization
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 518 | 528
mg/dL | 2.2 (0.1) | 2.1 (0.1)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.1]

14. Secondary Outcome: New Vasopressor Use to Day 7
Description: The number of subjects in each arm that are started on a vasopressor after randomization up to study day 7.
Time Frame: Up to 7 days after randomization
Population: need info on this
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 357 | 360
Participants | 43 | 42
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Risk Difference (RD) = 0.4, 95% CI 2-sided [-4.4 to 5.1]

15. Secondary Outcome: Highest Cardiovascular SOFA (Sepsis Related Organ Failure Assessment) Score
Description: Cardiovascular score of the Organ SOFA score was used:
  Score = 0: MAP* >= 70 mmHg and No Drug;
  Score = 1: MAP < 70 mmHg and No Drug;
  Score = 2: (Any MAP) ( dopamine<=5 OR any dobutamine ) AND no other drugs (include neosynephrine vasopressin);
  Score = 3: (Any MAP) 5 < dopamine <= 15 OR epinephrine <= 0.1 OR norepinephrine <= 0.1 OR neosynephrine <=0.22 OR any dose vasopressin;
  Score = 4: (Any MAP) dopamine > 15 OR epinephrine > 0.1 OR norepinephrine > 0.1 OR neosynephrine > 0.22
  * MAP = mean arterial pressure
Time Frame: Up to 7 days after randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 523 | 534
score on a scale | 1.4 (0.1) | 1.3 (0.1)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0]

16. Secondary Outcome: 25OHD Levels at Day 3
Description: Baseline levels will be measured using LC/MS/MS methods (all randomized participants) and at day 3 (the first 300 randomized participants only).
Time Frame: 3 days after randomization
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 145 | 133
ng/mL | 46.9 (23.2) | 11.4 (5.6)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 35.5, 95% CI 2-sided [31.5 to 39.6]

17. Secondary Outcome: Highest Total Calcium to Day 14
Description: Clinically available serum or ionized Ca levels were obtained through day 14 for all randomized patients. This time frame was selected to align with the 25OHD half life of two weeks.
Time Frame: 14 days after randomization
Population: Subjects with a clinically available total calcium level up to study day 14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 507 | 513
mg/dL | 8.9 (0.8) | 8.8 (0.7)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; p = 0.004, t-test, 2 sided

18. Secondary Outcome: Highest Ionized Calcium to Day 14
Description: Clinically available serum or ionized calcium levels through day 14 were collected for all randomized participants. This time frame was selected to align with the 25OHD half life of two weeks.
Time Frame: up to 14 days after randomization
Population: Subjects with a clinically available ionized calcium level up to study day 14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 153 | 177
mg/dL | 4.7 (0.8) | 4.6 (0.8)
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; p = 0.67, t-test, 2 sided

19. Secondary Outcome: Hypercalcemia to Day 14
Description: As the half-life of 25OHD is approximately 2 weeks, clinically available serum or ionized calcium levels through study day 14 were collected. The number of participants with hypercalcemia was reported.
Time Frame: up to 14 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 513 | 523
Participants | 14 | 11
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; p = 0.51, Chi-squared

20. Secondary Outcome: Kidney Stones to Day 90
Description: Incident of kidney stones determined by chart review at the end of hospitalization and by self-report at day 90 phone call in those discharged from the hospital prior to day 90.
Time Frame: 90 days after randomization
Population: Subjects discharged from the hospital prior to study day 90.
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 507 | 507
Participants | 0 | 3
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; p = 0.25, Fisher Exact

21. Secondary Outcome: Fall-related Fractures to Day 90
Description: Incident of fall-related fractures will be determined by chart review at the end of hospitalization and by self-report at day 90 phone call for those discharged from the hospital prior to day 90. Most data suggest that high dose vitamin D in healthy outpatients may improve muscle function, balance, and bone mineral density, and thus decrease fall-related fractures, but other data suggest that high dose vitamin D supplementation may actually increase the incidence of falls/fractures. Because of this uncertainty and limited data in hospitalized patients, we assessed for incident of fall-related fractures.
Time Frame: 90 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 507 | 507
Participants | 4 | 2
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; p = 0.69, Chi-squared

22. Secondary Outcome: Falls to Day 90
Description: We assessed for incidence of falls by chart review at the end of hospitalization and by self-report at the 90 day phone call. Most data suggest that high dose vitamin D in healthy outpatients may improve muscle function, balance, and bone mineral density, and thus decrease fall-related fractures, but other data suggest that high dose vitamin D supplementation may actually increase the incidence of falls/fractures.
Time Frame: 90 days post randomization
Population: need to give info
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Vitamin D Formulation | Placebo
Number analyzed (Participants) | 507 | 507
Participants | 36 | 27
Statistical Analysis 1: Comparison: High Dose Vitamin D Formulation vs Placebo; Test type: Superiority; p = 0.24, Chi-squared

ADVERSE EVENTS:
Time Frame: Subjects were assessed for adverse events from enrollment (signing of the informed consent) through study day 14 or hospital discharge, whichever occurs first. Investigators will determine if the event is serious or related to the study drug. The rationale for this time window is the 2 week half-life of 25OHD, which helps to define the period at risk from vitamin D.
Arm/Group | High Dose Vitamin D Formulation | Placebo
All-Cause Mortality (participants affected / at risk) | 159/681 | 137/656
Serious Adverse Events (participants affected / at risk) | 14/690 | 18/668
Other Adverse Events (participants affected / at risk) | 10/690 | 6/668
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D Formulation (N=690) | Placebo (N=668)
Altered Mental Status (Nervous system disorders) | 1 (1) | 1 (1)
Blindness (Nervous system disorders) | 0 (0) | 1 (1)
Breathing Kussmaul Type (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
C Difficile Toxin (Infections and infestations) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Colitis Pseudomembranous (Infections and infestations) | 0 (0) | 1 (1)
CVA (Nervous system disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
ED Visit (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fluid Overload (Cardiac disorders) | 0 (0) | 1 (1)
Hearing Impaired (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hemorrhage Jejunum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrahge Retroperitoneal (Vascular disorders) | 0 (0) | 1 (1)
Heparin Induced Thrombocytopenia and Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension, Unresponsive (Vascular disorders) | 1 (1) | 0 (0)
Lung Disease Obstructive (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PEA (Cardiac disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Cardiac disorders) | 0 (0) | 1 (2)
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Readmission (General disorders) | 2 (2) | 0 (0)
Readmission to MICU (General disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ureteral Calculus (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteral Obstruction from Renal Stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Weakness Left Sided (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vitamin D Formulation (N=690) | Placebo (N=668)
Anemia Microcytic (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Confidentiality (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Discoloration Urine (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea and Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypercalcemia (Endocrine disorders) | 2 (2) | 0 (0)
Platelets Decreased (Investigations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The Data and Safety Monitoring Board recommended that the trial be stopped at the first interim analysis when the primary outcome of the study crossed a protocol specified futility boundary. This adaptive design element resulted in a completed study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT03096314/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT03096314/SAP_001.pdf